CLINICAL TRIAL: NCT00108095
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Dose-ranging, Parallel Group Phase II Study to Evaluate the Safety, Efficacy and Pharmacokinetics of the Oral Neurokinin-1 Receptor Antagonist, GW679769, When Administered With Intravenous Ondansetron Hydrochloride for the Prevention of Post-operative Nausea and Vomiting (PONV) and Post-discharge Nausea and Vomiting (PDNV) in Female Subjects With Known Risk Factors for PONV Who Are Undergoing Surgical Procedures Associated With an Increased Emetogenic Risk
Brief Title: A Study To Evaluate An NK-1 Antiemetic For The Prevention Of Post Operative Nausea And Vomiting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NKT102260
Record Dates: First submitted 2005-04-13; First posted 2005-04-14 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Postoperative Nausea and Vomiting; Nausea and Vomiting, Postoperative
Keywords: emesis; nausea; post operative nausea and vomiting; vomiting; PONV
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Vomiting; Nausea

INTERVENTIONS:
Drug: intravenous ondansetron

SUMMARY:
This study is looking at a range of doses of this NK-1 receptor antagonist drug, for both safety and effectiveness in prevention PONV

DETAILED DESCRIPTION:
A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging, Parallel Group Phase II Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of the Oral Neurokinin-1 Receptor Antagonist, GW67969, When Administered With Intravenous Ondansetron Hydrochloride for the Prevention of Post-Operative Nausea and Vomiting (PONV) and Post-Discharge Nausea and Vomiting (PDNV) in Female Subjects With Known Risk Factors for PONV Who Are Undergoing Surgical Procedures Associated With an Increased Emetogenic Risk

ELIGIBILITY:
Inclusion criteria:

* Females age 18-55
* Laparoscopic/laparotomic gynecological procedure of laparoscopic gallbladder removal

Exclusion criteria:

* Pregnant or breastfeeding
* Post-menopausal
* Not undergoing general anesthesia

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 701 (Actual)
Dates: Start 2004-10; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Number of subjects who achieve a complete response (defined as no vomiting, no retching, no rescue therapy, and no premature discontinuation from the study) during the first 24 hour evaluation period following emergence from anesthesia

SECONDARY OUTCOMES:
Number of subjects who achieve a complete response during each subsequent 24 hour evaluation period (up to 120 hours)following the emergence from anesthesia
The extent of nausea experienced by subjects.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (53):
- United States (27):
  - GSK Investigational Site, Montgomery, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Arcadia, California
  - GSK Investigational Site, Duarte, California
  - GSK Investigational Site, Glendale, California
  - GSK Investigational Site, Laguna Hills, California
  - GSK Investigational Site, Loma Linda, California
  - GSK Investigational Site, Pasadena, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Stanford, California
  - GSK Investigational Site, Naples, Florida
  - GSK Investigational Site, Pensacola, Florida
  - GSK Investigational Site, Alpharetta, Georgia
  - GSK Investigational Site, Hutchinson, Kansas
  - GSK Investigational Site, Kansas City, Kansas
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, New Brunswick, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Winchester, Virginia
  - GSK Investigational Site, Wenatchee, Washington
- Belgium (3):
  - GSK Investigational Site, Aalst
  - GSK Investigational Site, Braasschaat
  - GSK Investigational Site, Brussels
- Canada (12):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Ste-Foy, Quebec
- Germany (3):
  - GSK Investigational Site, Marburg, Hesse
  - GSK Investigational Site, Aachen, North Rhine-Westphalia
  - GSK Investigational Site, Koblenz, Rhineland-Palatinate
- Hungary (4):
  - GSK Investigational Site, Győr
  - GSK Investigational Site, Kistarcsa
  - GSK Investigational Site, Miskolc
  - GSK Investigational Site, Székesfehérvár
- Spain (4):
  - GSK Investigational Site, Cadiz
  - GSK Investigational Site, Cartagena
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Santiago de Compostela

REFERENCES:
- [Background] Singla NK, Singla SK, Chung F, Kutsogiannis DJ, Blackburn L, Lane SR, Levin J, Johnson B, Pergolizzi JV Jr. Phase II study to evaluate the safety and efficacy of the oral neurokinin-1 receptor antagonist casopitant (GW679769) administered with ondansetron for the prevention of postoperative and postdischarge nausea and vomiting in high-risk patients. Anesthesiology. 2010 Jul;113(1):74-82. doi: 10.1097/ALN.0b013e3181d7b13a. PMID 20526194